CLINICAL TRIAL: NCT05475366
Title: Pilot Study of Personalized First-line Chemotherapy Choice for Patients With Advanced Pancreatic Adenocarcinoma Using Transcriptomic Signatures (PACsign)
Brief Title: Personalized First-line Chemotherapy Choice in Advanced Pancreatic Adenocarcinoma Using Transcriptomic Signatures (PACsign)
Acronym: PACsign
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2021-15
Record Dates: First submitted 2022-07-07; First posted 2022-07-26 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma, Pancreatic Ductal; Prognosis
Keywords: Transcriptomic signatures; Personalized first-line chemotherapy; Metastatic PDAC
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Anophthalmia with pulmonary hypoplasia | interventions — Long Interspersed Nucleotide Elements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Molecular screening for prediction of response (Experimental): L1 chemotherapy regimen (FOLFIRINOX vs Gemcitabine plus nab-paclitaxel (GemnabP)) will be selected based on transcriptomic signatures applied to the pre-therapeutic biopsy of newly diagnosed PDAC patients.
  Interventions: Other: Clinical value of 5 transcriptomic signatures to personalize the therapeutic decision for L1 in PDAC; Other: Biomarkers of tumor signatures (translational studies)

INTERVENTIONS:
Other: Clinical value of 5 transcriptomic signatures to personalize the therapeutic decision for L1 in PDAC — Formalin-Fixed Paraffin-Embedded (FFPE) samples will be centralized in which nucleic acids extraction (DNA+RNA) and FFPE-compatible RNA-sequencing will be performed in real-time (≤28 days). RNAseq reads will be processed and all 5 transcriptomic signatures will be applied for prediction of response to 5FU, oxaliplatin, irinotecan, gemcitabine and taxane. In addition, biomarkers status will be obtained for all patients as part of good clinical practice.
Other: Biomarkers of tumor signatures (translational studies) — Blood (serum and plasma) will be drawn at baseline, week 8, and tumor progression in order to look for surrogate biomarkers of tumor signatures in liquid biopsy

SUMMARY:
The aim of this study is to assess the clinical value of 5 transcriptomic signatures prognostic of chemotherapeutic sensitivity to improve the Objective Response Rate (ORR) of first-line (L1). Chemotherapy regimen (FOLFIRINOX vs Gem-nabP) will be selected based on transcriptomic signatures applied to the pre-therapeutic liver biopsy of newly diagnosed PDAC patients.

DETAILED DESCRIPTION:
Step 1: patients will sign a 1st informed consent prospectively for the molecular screening (RNAseq profile). 5 transcriptomic signatures will be applied for prediction of response to 5 Fluoro-Uracil (5FU), oxaliplatin, irinotecan, gemcitabine and taxane. Biomarker status will be obtained for all patients as part of good clinical practice.

Patients will be eligible for prospective step 2 only if the transcriptomic analysis is informative and the treatment can be started within 28 days.

Step 2: study treatment strategy: based on the results of transcriptomic signatures, patients will receive either FOLFIRINOX or Gem-nabP according to the following algorithm (2nd informed consent):

* Predicted to be FOLFIRINOX sensitive (regardless of sensitivity to Gem-nabP) = FOLFIRINOX
* Predicted to be FOLFIRINOX and Gem-nabP resistant = FOLFIRINOX
* Presence of a germline breast cancer (BRCA) mutation (regardless of transcriptomic signature) = FOLFIRINOX (tumors sensitive to platinum).
* Predicted to be Gem-nabP sensitive and FOLFIRINOX resistant = Gem-nabP

Chemotherapy with FOLFIRINOX and Gemcitabine plus nab-paclitaxel will be administered as in routine practice, according to their approval. Dose adaptation will be allowed according to investigator's usual practice.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.
2. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
3. Histologically or cytologically proven Pancreatic Ductal Adenocarcinoma (PDAC).
4. Metastatic disease.
5. Measurable or evaluable lesions according to RECIST v1.1 criteria.
6. First-line therapy (previous neoadjuvant/adjuvant chemotherapy not allowed).
7. Age ≥ 18 years (no upper limit, patients ≥ 75 years old must have a G8 score ≥ 14).
8. 3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1.
9. Availability of tumor tissue sample from the primary pancreatic tumor or liver metastasis (chemo-naïve) before inclusion in step 1.
10. Adequate organ function, as defined by the following (blood test ≤ 7 days prior to inclusion):

    1. Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN) (≤ 5 ULN in case of liver metastases)
    2. Total serum bilirubin ≤ 1.5 ULN
    3. Serum albumin ≥ 28 g/L
    4. Hemoglobin ≥ 9.0 g/dl
    5. Absolute neutrophil count (ANC) ≥ 1,500/μL
    6. Platelets ≥ 100,000/μL
    7. Creatinine clearance ≥ 50 mL/min (MDRD).
11. No Dihydropyrimidine dehydrogenase (DPD) deficiency (normal uracil level).
12. Life expectancy ≥ 3 months.
13. a. Evidence of post-menopausal status b. (or) negative urinary or serum pregnancy test for female pre-menopausal patients.
14. Registration in a National Health Care System.

Exclusion Criteria:

1. Concurrent enrolment in another interventional clinical study.
2. Previous treatment with chemotherapy for pancreatic cancer.
3. Uncontrolled massive pleural effusion or massive ascites.
4. Known deficiency in UGT1A1 (homozygous UGT1A1*28 allele).
5. Active bacterial, viral, or fungal infection requiring systemic therapy, including tuberculosis, hepatitis B (known positive Hepatitis B Virus surface antigen (HBsAg) result), hepatitis C (with positive RNA), Sars-Cov-2 or human immunodeficiency virus (positive HIV 1/2 antibodies).
6. Diagnosis of any second malignancy within the last 3 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri.
7. Known active central nervous system metastases and/or carcinomatous meningitis; patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline).
8. Uncontrolled intercurrent illness, including but not limited to, symptomatic congestive heart failure or coronary disease, peripheral artery disease, severe chronic obstructive pulmonary disease, decompensated cirrhosis, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
9. Live vaccine administration within 30 days prior to the first dose of study treatment.
10. Known or suspected allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
11. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with participation for the full duration of the trial, or is not in the best interest of the participant, in the opinion of the treating investigator.
12. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
13. Major surgical procedure (as defined by the Investigator) within 4 weeks prior to the first dose of trial treatment.
14. Pregnancy/lactation.
15. Person under legal protection or tutelage or guardianship.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2028-12-11 (Estimated); Study Completion 2028-12-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) at 4 months based on thorax-abdomen-pelvis (TAP) CT scan every 8 weeks according to RECIST v1.1. | 4 months
  ORR, defined as the percentage of patients whose disease decreased by at least 30% (partial response - PR) and/or disappeared (complete response - CR) under treatment among patients who start treatment.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 18 months
  PFS, defined as the time from the date of treatment initiation to the date of progression or death whatever the cause. Progression will be assessed by the investigator based on TAP-CT scan every 8 weeks according to RECIST v1.1.
Overall Survival (OS) | 18 months
  OS, defined from the date of treatment initiation to the date of death whatever the cause.
Disease Control Rate (DCR) | 18 months
  DCR, defined as the percentage of patients who have achieved complete response, partial response or stable disease according to RECIST v1.1 among patients who start treatment.
Treatment-related severe (grade 3-5) toxicities | 18 months
  Toxicities will be graded, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (digestive, hematologic, neuropathy).
Feasibility of study procedure | 12 months
  Measured as the rate of usable samples

CONTACTS AND LOCATIONS:
Overall Officials: Cindy NEUZILLET, MD, PhD, Study Director — Institut Curie
Locations (6):
- France (6):
  - Hôpital Beaujon, Clichy
  - Hôpital HENRI MONDOR, Créteil
  - Hôpital Claude Hurriez, Lille
  - Institut Paoli-Calmettes, Marseille
  - CHU Robert Debré, Reims
  - Institut Curie, Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).